CLINICAL TRIAL: NCT07043569
Title: Clinical-randomized Trial of the Effect of Rehabilitation Therapy Using Strength and Blood Flow Restriction Training on Muscular Fitness and Regeneration After Anterior Cruciate Ligament Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Alexander Franz, Dr. med., B.Sc., University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024_F
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-06

CONDITIONS: ACL - Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Control group will perform the exercise protocols with a sham-BFR pressure of 20 mmHg.
  Interventions: Other: Resistance Training with Sham-BFR
- Intervention Group (Experimental): Intervention group will perform the exercise protocols with a BFR pressure corresponding to 60% of the individual limb occlusion pressure.
  Interventions: Other: Resistance Exercise with BFR

INTERVENTIONS:
Other: Resistance Training with Sham-BFR — The exercise protocol provides for units of approx. 25 minutes of BFR training five times a week as part of medical training therapy. Based on the initial strength measurements prior to rehabilitation, the training phase of the intervention group starts with 30% of the 1RM (calculated from the force-velocity profile) and 70% LOP in the operated leg and 75% of the 1RM (calculated from the force-velocity profile) in the unoperated leg. The patients are randomized into 2 groups: 1) intervention group, which receives a daily intervention with an occlusion pressure and the 2) control group, which receives a daily "Sham-BFR" intervention with an occlusion pressure of 20mmHg.
  Arms: Control Group
Other: Resistance Exercise with BFR — The exercise protocol provides for units of approx. 25 minutes of BFR training five times a week as part of medical training therapy. Based on the initial strength measurements prior to rehabilitation, the training phase of the intervention group starts with 30% of the 1RM (calculated from the force-velocity profile) and 70% LOP in the operated leg and 75% of the 1RM (calculated from the force-velocity profile) in the unoperated leg. The patients are randomized into 2 groups: 1) intervention group, which receives a daily intervention with an occlusion pressure and the 2) control group, which receives a daily "Sham-BFR" intervention with an occlusion pressure of 20mmHg.
  Arms: Intervention Group

SUMMARY:
With the intention of improving rehabilitation after anterior cruciate ligament reconstruction, the present project investigates the influence of a targeted strength and blood flow restriction training intervention (BFR training) on the regeneration of muscle mass, strength and functionality of the knee joint. BFR training is characterized by the combination of external venous vascular occlusion with light strength training and still enables users to achieve gains in muscle mass and strength that are comparable to training with high mechanical loads. The positive effects of BFR training in the course of knee arthroplasty have already been demonstrated by our working group as a prehabilitative approach, i.e. as a training intervention prior to surgery. In the present project, the framework conditions of outpatient rehabilitation at the Bonn Center for Outpatient Rehabilitation will now be used to prove whether sports science-controlled strength and BFR training has a similar effect in the postoperative rehabilitation phase. The interventions are carried out as part of the exercise therapy units in outpatient rehabilitation ETM01 in accordance with the S2k guideline on anterior cruciate ligament rupture. Strength and BFR training in medical training therapy supplements the daily exercise therapy to ensure implementation in the rehabilitation process in line with the guidelines.

ELIGIBILITY:
Inclusion Criteria:

* ACL reconstruction
* Ability to take part in an outpatient rehabilitation

Exclusion Criteria:

* Sickle Cell anemia
* iatrogenic changes in the vessels of the lower limbs (stents, bypasses)
* inflammation of the lower extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle Strength (N) | Pre- (before Rehabilitation) to Post-Rehabilitation (immediately after three weeks of exercise intervention up to 1 year follow up)
  isoemtric maximal strength of both legs will assessed on a isokinetic leg press.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No